CLINICAL TRIAL: NCT02968810
Title: Statin Therapy to Reduce Disease Progression From Liver Cirrhosis to Cancer
Brief Title: Simvastatin in Preventing Liver Cancer in Patients With Liver Cirrhosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2016-01719; NCI-2016-01719 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00035; NCI2015-06-03 (Other: Northwestern University); NWU2015-06-03 (Other: DCP); N01CN00035 (NIH); P30CA060553 (NIH)
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Results first posted 2025-04-15 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-06

CONDITIONS: Cirrhosis; Hepatocellular Carcinoma
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (simvastatin) (Experimental): Patients receive simvastatin PO QD. Treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood on study and CT/MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Drug: Simvastatin
- Group II (placebo) (Placebo Comparator): Patients receive placebo PO QD. Treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood on study and CT/MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Placebo Administration — Given PO
  Arms: Group II (placebo)
Other: Questionnaire Administration — Ancillary studies
Drug: Simvastatin — Given PO
  Other Names: MK 733; Synvinolin; Zocor
  Arms: Group I (simvastatin)

SUMMARY:
This phase II trial studies how well simvastatin works in preventing liver cancer in patients with liver cirrhosis. Simvastatin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of a simvastatin intervention versus placebo on the change in serum AFP-L3% from baseline to 6 months following treatment initiation in patients with liver cirrhosis who have a current model for end-stage liver disease (MELD) =< 20.

SECONDARY OBJECTIVES:

I. To evaluate the effect of a simvastatin intervention versus placebo at 6 months from baseline on the change in:

Ia. Serum AFP; Ib. Serum IL-6; Ic. Serum deoxycholic acid; Id. Liver stiffness; Ie. Fibrosis 4 index (FIB-4) score; If. MELD score.

EXPLORATORY OBJECTIVES:

I. To evaluate the effect of a simvastatin intervention versus placebo at 6 months from baseline on the change in other:

Ia. serum bile acid levels; Ib. serum immune markers.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive simvastatin orally (PO) once daily (QD). Patients also undergo collection of blood on study and computed tomography (CT) scans/magnetic resonance imaging (MRI) throughout the trial.

GROUP II: Patients receive placebo PO QD. Patients also undergo collection of blood on study and CT/MRI throughout the trial.

In both groups, treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30, 60, and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of liver cirrhosis assessed by the presence of clinical signs, symptoms, body imaging (ultrasound, computed tomography [CT], or magnetic resonance imaging [MRI]), or liver biopsy
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 2,500/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 50,000/microliter
* Hemoglobin >= 8 g/dL
* Total bilirubin =< 3 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 x institutional ULN
* Creatinine =< 1.5 x institutional ULN
* Women who are able to become pregnant must have a confirmed negative pregnancy test result prior to enrollment; women >= 50 years of age who have not had a menstrual period in the past year; and women who have had a hysterectomy, both ovaries removed, or a tubal ligation; will not be required to have a pregnancy test
* The effects of simvastatin on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women who are able to become pregnant must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document and medical release
* Willing and able to comply with trial protocol and follow-up
* Have had an abdominal imaging test (CT, MRI, or ultrasound) within the past 18 months

Exclusion Criteria:

* Prior or current use of statin medication
* Current systemic use of medications known to interact with statins and potentially increase toxicity, including gemfibrozil, cyclosporine, danazol, lomitapide, verapamil, diltiazem, dronedarone, amiodarone, amlodipine, ranolazine, strong CYP3A4 inhibitors (e.g., itraconazole, ketoconazole, posaconazole, voriconazole, human immunodeficiency virus [HIV] protease inhibitors, boceprevir, telaprevir, erythromycin, clarithromycin, telithromycin, nefazodone, or cobicistat-containing products), or strong CYP3A4 inducers (e.g., carbamazepine, phenytoin, rifampin, St. John's wort, bosentan, efavirenz, etravirine, modafinil, nafcillin)
* History of adverse effects, intolerance, or allergic reactions attributed to compounds of similar chemical or biologic composition to simvastatin (i.e., other statin medications)
* Current use of any other investigational agents
* Women who are pregnant or breastfeeding; pregnant women are excluded from this study because simvastatin is a lipid-lowering agent with the potential for teratogenic or abortifacient effects; it is not known whether simvastatin is excreted into human milk; however, a small amount of another drug in this class does pass into breast milk; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with simvastatin, breastfeeding should be discontinued if the mother is treated with simvastatin
* Prior liver transplant
* Prior known or suspected hepatocellular carcinoma
* Prior cholangiocarcinoma
* Model for end-stage liver disease (MELD) > 20
* Any lab results that do not meet inclusion criteria after the Screen 1 blood tests
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of chronic myopathy
* Prior germ cell cancer
* History of active malignancy within the past 5 years (excluding basal/squamous cell skin cancer or prostate cancer with a Gleason score 6 or less)
* Known active infection with HIV
* Medical contraindications to blood draw (e.g., hemophilia)
* Concurrent illness which in the opinion of the investigators would compromise either the patient or the integrity of the data
* Current excessive alcohol consumption (average alcohol consumption of more than 5 drinks per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2025-12-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marc T Goodman, Principal Investigator — Northwestern University
Locations (5):
- United States (3):
  - Cedars Sinai Medical Center, Los Angeles, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
- Puerto Rico (2):
  - Centro Comprensivo de Cancer de UPR, San Juan
  - University of Puerto Rico, San Juan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 59 participants were randomized. 52 out of 59 participants started study agent.
Groups:
- Group I (Simvastatin): Patients receive simvastatin PO QD. Treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity.
- Group II (Placebo): Patients receive placebo PO QD. Treatment continues for up to 6 months in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Group I (Simvastatin) | Group II (Placebo)
Started | 28 | 24
Completed | 25 | 20
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Disease Progression | 0 | 1

BASELINE CHARACTERISTICS:
Population: 59 participants were randomized. 52 out of 59 participants started study agent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Simvastatin) | Group II (Placebo) | Total
Number analyzed (Participants) | 28 | 24 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9.0) | 59 (7.4) | 59 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 17 | 13 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 15 | 11 | 26
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 24 | 19 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 4 | 3 | 7
  United States | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum AFP-L3%
Description: Assessed by liquid-phase binding assay. Mean AFP-L3% difference calculated including all participants imputing undetectable values with 0.5%
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Group I (Simvastatin) | Group II (Placebo)
Number analyzed (Participants) | 25 | 20
percent | 0.24 (1.00) | -0.04 (0.11)

2. Secondary Outcome: Change in Serum AFP
Description: Assessed by liquid-phase binding assay. Mean difference in AFP, a glycoform produced by malignant liver cells.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Group I (Simvastatin) | Group II (Placebo)
Number analyzed (Participants) | 25 | 20
ng/ml | .39 (1.33) | -0.09 (0.4)

3. Secondary Outcome: Change in Serum IL-6
Description: Mean difference in IL-6 (interleukin-6) NPX (normalized protein expression).
Time Frame: Baseline to 6 months
Measure: Mean (Inter-Quartile Range); unit: normalized protein expression
Arm/Group | Group I (Simvastatin) | Group II (Placebo)
Number analyzed (Participants) | 25 | 20
normalized protein expression | -0.49 [-1.39 to 0.15] | 0.25 [-0.31 to 0.48]

4. Secondary Outcome: Change in Serum Deoxycholic Acid
Description: Assessed by liquid chromatography coupled with mass spectrometry. Median difference in serum DCA (deoxycholic acid), a secondary bile acid.
Time Frame: Baseline to 6 months
Measure: Median (Inter-Quartile Range); unit: pmol/gram
Arm/Group | Group I (Simvastatin) | Group II (Placebo)
Number analyzed (Participants) | 25 | 20
pmol/gram | 0.00 [-60.0 to 55.3] | 0.00 [-68.0 to 4.89]

5. Secondary Outcome: Change in Liver Stiffness
Description: Assessed by liver elastography. Fibroscan score from a fibroscan examination (a non-invasive measurement of liver fibrosis). A test result of greater than 20kPa is generally associated with an increased HCC risk. Mean difference in liver stiffness.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: kPA
Arm/Group | Group I (Simvastatin) | Group II (Placebo)
Number analyzed (Participants) | 25 | 20
kPA | 3.89 (15) | 3.83 (14.1)

6. Secondary Outcome: Change in Fibrosis 4 Index Score
Description: The Fib-4 index is a non-invasive measure of liver stiffness. A high score (FIB4 ≥ 3.25) and low score is (FIB4 < 1.3) The FIB-4 index is calculated as follows: FIB-4 = (Age × AST (U/L)) ÷ (PLT (109/L) × (√ ALT (U/L)). Change in mean difference.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (Simvastatin) | Group II (Placebo)
Number analyzed (Participants) | 25 | 20
score on a scale | 0.4 (1.20) | 0.17 (1.22)

7. Secondary Outcome: Change in Model for End-Stage Liver Disease Score
Description: The Model for End-Stage Liver Disease (MELD) is a validated predictor of survival among different populations of patients with advanced liver disease. MELD = 9.57 x ln(creatinine [mg/dL]) + 3.78 x ln(total bilirubin [mg/dL]) + 11.2 x ln(INR) + 6.43. Scores range from 6 (low/ less liver disease) to 40 (high/severe liver disease). Change in mean difference.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (Simvastatin) | Group II (Placebo)
Number analyzed (Participants) | 25 | 20
score on a scale | 0.57 (2.76) | 0.18 (1.61)

ADVERSE EVENTS:
Time Frame: Collected from the time informed consent was signed and baseline procedures were completed through 90 days post-intervention.
Arm/Group | Group I (Simvastatin) | Group II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/24
Serious Adverse Events (participants affected / at risk) | 3/28 | 3/24
Other Adverse Events (participants affected / at risk) | 24/28 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Simvastatin) (N=28) | Group II (Placebo) (N=24)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) — Sepsis
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) — Infection/septic shock
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) — Calculus
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Noninvasive tonsil cancer
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Simvastatin) (N=28) | Group II (Placebo) (N=24)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal disorders - Other, specify (inguinal hernia) (Gastrointestinal disorders) | 2 (2) | 0 (0) — Acid reflux
Fatigue (General disorders) | 0 (0) | 6 (6)
Flu like symptoms (General disorders) | 4 (4) | 4 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (4) | 2 (2)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 6 (16) | 6 (12)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT02968810/Prot_SAP_000.pdf